CLINICAL TRIAL: NCT06991101
Title: Randomized Phase 2 Trial of Ruxolitinib in Combination With Radiation and Temozolomide Compared to Radiation and Temozolomide for Newly Diagnosed Glioblastoma.
Brief Title: Ruxolitinib With Radiation and Temozolomide Compared to Radiation and Temozolomide for Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-AHL-001
Record Dates: First submitted 2025-05-19; First posted 2025-05-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma; Brain Cancer; Glioblastoma Multiforme; Glioblastoma Multiforme of Brain; Glioblastoma Multiforme, Adult; MGMT-Unmethylated Glioblastoma; MGMT-Methylated Glioblastoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — ruxolitinib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib plus Radiation and Temozolomide (Experimental): There will be two phases of drug administration: (1) Ruxolitinib and temozolomide will be administered "During Radiation Therapy" and (2) Maintenance phase after radiation therapy is complete.
  Interventions: Drug: Ruxolitinib; Drug: Temozolomide; Radiation: Radiation Therapy
- Radiation and Temozolomide (Active Comparator): There will be two phases of drug administration: (1) Temozolomide will be administered "During Radiation Therapy" and (2) Maintenance phase after radiation therapy is complete.
  Interventions: Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Ruxolitinib — "During Radiation Therapy" phase: 20 mg ruxolitinib will be self-administered orally (PO) twice every day (BID), starting on Day 1 for 6 weeks. Then there will be a 4-week break after radiotherapy is complete.
  "Maintenance" phase: Occurs thirty days (4 weeks) after receiving the last dose of radiotherapy. Ruxolitinib 20 mg will be self-administered PO BID, starting on Day 1 in consecutive 28-day cycles.
  Either phase:
  Aside from the 30-day break, ruxolitinib will be continued daily until disease progression or treatment intolerance. Ruxolitinib should be administered at approximately the same time each day. The tablets should be swallowed whole with water and should not be opened, broken, or chewed. The dose may be reduced in the case of certain adverse events.
  Other Names: Jakavi
  Arms: Ruxolitinib plus Radiation and Temozolomide
Drug: Temozolomide — "During Radiation Therapy" phase: 75 mg/m^2 will be self-administered PO once every day, starting on Day 1, for 6 weeks. Then there will be a 4-week break after radiotherapy is complete.
  "Maintenance" phase: Occurs thirty days (4 weeks) after receiving the last dose of radiotherapy. Temozolomide 150-200 mg/m^2 will be self-administered PO BID, starting on Day 1 to Day 5 of each cycle for six cycles.
  Either phase:
  The dose may be reduced in the case of certain adverse events.
  Other Names: Temodar
Radiation: Radiation Therapy — Radiation will be administered every weekday (Monday to Friday) in 2 Gy fractions for 30 fractions during a 6-week period (60 Gy total).

SUMMARY:
The purpose of this research is to test the safety and effectiveness of the investigational drug ruxolitinib when it is combined with standard of care treatment (radiation therapy and temozolomide) for the treatment of newly diagnosed glioblastoma. Half the people in the study will be assigned to take the study drug ruxolitinib in addition to the standard of care temozolomide and radiation therapy and the other half will be assigned to the standard of care temozolomide and radiation therapy only. This assignment will be randomized in a 1-to-1 ratio, like the flip of a coin.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Individuals of any sex, gender, race, or ethnicity ≥ 18 years of age.
4. Histologically confirmed glioblastoma as defined by the World Health Organization (WHO) 2021 Criteria (IDH-wildtype) that is either methylated, unmethylated, or indeterminate MGMT.
5. Confirmation that patient has sufficient tissue to undergo MGMT and IDH testing, as mandated.
6. Must have a Karnofsky performance status (KPS) ≥ 70% (i.e., the patient must be able to care for themself with occasional help from others).
7. Adequate organ (liver and renal) and bone marrow function within 14 days before randomization. For all parameters listed below, the most recent results available must be used:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3. Note: Granulocyte-colony stimulating factor (G-CSF) administration is not allowed within 1 week prior to screening assessment.
   2. Platelet count ≥ 100,000/mm3. Note: Platelet transfusion is not allowed within 1 week prior to registration.
   3. Total bilirubin (TBL) ≤ 1.5 × institutional upper limit of normal (ULN).
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.
   5. Serum albumin ≥ 2.5 g/dL.
8. Patients able to become pregnant: use of highly effective contraception for at least one (1) month prior to screening and agreement to use such a method. Should a participant become pregnant or suspect that they are pregnant while participating in this study, they should notify the treating physician immediately. Such individuals must have a negative pregnancy test.
9. Patients must have no concurrent malignancy except curatively treated early-stage bladder and prostate cancer that has been completed resected, basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission. Patients with other prior malignancies must be disease-free for ≥ 3 years.

Exclusion Criteria:

1. Patients who are pregnant or breast-feeding. The anti-proliferative activity of this experimental drug and temozolomide may be harmful to the developing fetus or nursing infant.
2. Patients receiving concurrent therapy for their brain tumor (e.g., chemotherapeutics or investigational agents).
3. Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for at least 3 years are eligible for this study.
4. Patients who have had repeat craniotomy for tumor therapy after receiving radiation therapy and temozolomide treatment.
5. Patients who received other chemotherapeutics or investigational agents in addition to their radiation therapy and concomitant temozolomide treatment.
6. Patient has previously taken ruxolitinib or is allergic to components of the study drug.
7. Patients using warfarin.
8. Uncontrolled immunodeficiency virus infection or active tuberculosis.
9. Patients with active serious infections requiring systemic therapy.
10. Known Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Participants with previous positive serology results must have negative polymerase chain reaction results.
11. Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, New York Heart Association (NYHA) Grade ≥2 heart failure, uncontrolled hypertension, valvular disease, pericarditis, myocardial infarction, or other thrombosis events like including pulmonary embolism or deep vein thrombosis within 6 months of screening.
12. Any other serious medical/psychiatric condition, in the judgement of the investigator, that likely to interfere or limit compliance with study requirements/treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) at end of study | 4 years
  OS is defined as the time from first treatment until the date of death from any cause at the end of the study. Participants who are lost to follow-up will be censored at the time of the last follow-up.

SECONDARY OUTCOMES:
OS at 12 months | 12 months
  OS is defined as the time from first treatment until the date of death from any cause at 12 months. Participants who are lost to follow-up will be censored at the time of the last follow-up.
Progression-free survival (PFS) at 6 months | 6 months
  PFS is defined as defined as the time from allocation to the first documented progressive disease (PD) using modified Response Assessment in Neuro-Oncology (mRANO) criteria or death due to any cause, whichever occurs first by 6 months. Participants who are lost to follow-up will be censored at the time of the last follow-up. PD is defined as any of the following events: 25% or more increase in sum of products of perpendicular diameters or ≥ 40% increase in total volume of enhancing lesions compared to the smallest tumor measurement obtained either at baseline or best response and sustained for at least 4 weeks; any new measurable (> 10mm × 10mm) enhancing lesions if baseline or best response demonstrated no measurable enhancing disease; clear clinical deterioration not attributable to other causes apart from tumor; or failure to return for evaluation as a result of death or deteriorating condition.
PFS at 12 months | 12 months
  PFS is defined as defined as the time from allocation to the first documented PD using mRANO criteria or death due to any cause, whichever occurs first by 12 months. Participants who are lost to follow-up will be censored at the time of the last follow-up. PD is defined above for PFS at 6 months.
Objective response rate (ORR) | 4 years
  ORR is defined as the proportion of participants in the analysis population who have a complete or partial response (CR or PR) using modified Response Assessment in Neuro-Oncology (mRANO) criteria. CR is defined as the disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks, no new lesions, stable or better neurological status, and no steroid use. PR is defined as 50% or more decrease in the in sum of the products of perpendicular diameters of all lesions or 65% or more decrease in total volume of all measurable enhancing lesions compared with baseline, sustained for at least 4 weeks, steroid use should be the same or lower compared to baseline, and neurological status should be stable or better compared to baseline.
Duration of response (DOR) | 4 years
  DOR is defined as the time that criteria for CR or PR (whichever is recorded first) is met until the date that recurrent or PD is objectively documented or expiration. mRANO will be used to assess response. PD is defined above for PFS at 6 months. CR and PR are defined above for ORR.
Incidence of Adverse Events (AEs) | 4 years
  An AE is defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered to be intervention-related. AEs will be documented from the time that the informed consent form is signed to the end of participation on the study. The number of total AEs will be calculated for this outcome.
Incidence of Serious Adverse Events (SAEs) | 4 years
  An SAE is defined as an AE that results in any of the following outcomes:
  * Death
  * Life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Congenital anomaly/birth defect
  Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  SAEs will be documented from the time that the informed consent form is signed to the end of participation on the study. The number of total SAEs will be calculated for this outcome.
Mortality | 4 years
  Number of participants who expire while on study.
Incidence of laboratory abnormalities | 4 years
  Laboratory values that fall outside the normal range will be documented, whether or not the values are considered clinically significant. The number of total laboratory abnormalities will be calculated for this outcome.
  Note: clinically significant laboratory abnormalities also will be documented as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, M.D., MBA, Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Ostrom QT, Kruchko C, Patil N, Tihan T, Cioffi G, Fuchs HE, Waite KA, Jemal A, Siegel RL, Barnholtz-Sloan JS. Brain and other central nervous system tumor statistics, 2021. CA Cancer J Clin. 2021 Sep;71(5):381-406. doi: 10.3322/caac.21693. Epub 2021 Aug 24. PMID 34427324
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Cao Y, Lathia JD, Eyler CE, Wu Q, Li Z, Wang H, McLendon RE, Hjelmeland AB, Rich JN. Erythropoietin Receptor Signaling Through STAT3 Is Required For Glioma Stem Cell Maintenance. Genes Cancer. 2010 Jan 1;1(1):50-61. doi: 10.1177/1947601909356352. PMID 20657792
- [Background] Guryanova OA, Wu Q, Cheng L, Lathia JD, Huang Z, Yang J, MacSwords J, Eyler CE, McLendon RE, Heddleston JM, Shou W, Hambardzumyan D, Lee J, Hjelmeland AB, Sloan AE, Bredel M, Stark GR, Rich JN, Bao S. Nonreceptor tyrosine kinase BMX maintains self-renewal and tumorigenic potential of glioblastoma stem cells by activating STAT3. Cancer Cell. 2011 Apr 12;19(4):498-511. doi: 10.1016/j.ccr.2011.03.004. PMID 21481791
- [Background] Becker H, Engelhardt M, von Bubnoff N, Wasch R. Ruxolitinib. Recent Results Cancer Res. 2014;201:249-57. doi: 10.1007/978-3-642-54490-3_16. PMID 24756798
- See also: Miami Cancer Institute — https://baptisthealth.net/services/cancer-care/miami-cancer-institute